CLINICAL TRIAL: NCT01107860
Title: Cone Beam Computed Tomography for Breast Imaging
Status: Completed | Type: Observational
Sponsor: Koning Corporation (Industry)
Collaborators: Elizabeth Wende Breast Care, LLC (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: KBCT-003; 2R44CA103236-05A1 (NIH)
Record Dates: First submitted 2010-01-05; First posted 2010-04-21 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group I
  Interventions: Device: Computed Tomography
- Group II
  Interventions: Device: Computed Tomography

INTERVENTIONS:
Device: Computed Tomography — In Group I, fifty CBCT studies will be performed. The objectives will be to illustrate the capacity of CBCT to image the breast in its entirety as compared with the gold standard mammographic exam.
  Groups: Group I
Device: Computed Tomography — In Group II , at least three hundred and fifty (350) study participants, who require diagnostic evaluation of the breast will undergo a breast CBCT . These subjects may be referred for biopsy as a result of a finding from a mammogram, ultrasound, MRI, or clinical exam.
  Groups: Group II

SUMMARY:
The primary aim of this study is to continue the investigation of cone beam computed tomography (CBCT) for breast imaging already underway in the diagnostic setting by providing a compelling body of evidence incorporating non-contrast CBCT in the study protocol. The goal is to accumulate a body of evidence to provide data to incorporate CBCT into the diagnostic work-up of breast lesions.

ELIGIBILITY:
Inclusion Criteria:

Group I:

* Females at least 35 years of age of any ethnicity
* Had a mammogram, read as BI-RADS® 1 or 2
* Will undergo study imaging no later than four weeks from date of mammogram.
* Is able to undergo informed consent.

Group II:

* Females at least 35 years of age of any ethnicity
* Require diagnostic imaging
* Will undergo study imaging no later than four weeks from date of diagnostic mammogram
* Is able to undergo informed consent

Exclusion Criteria:

Group I and Group II:

* Pregnancy
* Lactation
* Subjects with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Subjects who are unable to tolerate study constraints.
* Subjects who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to)

  * Treatment for enlarged thymus gland as an infant
  * Irradiation for benign breast conditions, including breast inflammation after giving birth
  * Treatment for Hodgkins disease
* Subjects who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Subjects who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to)

  * Tuberculosis
  * Severe scoliosis

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from the patient population at a community based clinic, Elizabeth Wende Breast Care, LLC, which is located in Rochester, NY. Group I will consist of subjects who have had mammograms read as BIRADS® 1 or 2. Group II will be subjects who have had a diagnostic mammogram read as BIRADS® 4 or 5 prior to breast biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Concordance and discordance of CBCT imaging with diagnostic mammography, other breast-imaging modalities, and histopathology | about 3 years
  The primary measure of this study will include the following aspects.
  * the capacity of CBCT to image the breast in its entirety as compared with the gold standard mammographic exam
  * patient's comfort during the CBCT exam vs the mammographic exam
  * the concordance and discordance of CBCT breast imaging with standard mammography and other breast-imaging studies
  * the concordance and discordance of CBCT breast imaging with histopathology
  * number of participants with adverse events as a measure of safety

CONTACTS AND LOCATIONS:
Overall Officials: Posy Seifert, D.O., Principal Investigator — Elizabeth Wende Breast Care, LLC
Locations (1):
- Elizabeth Wende Breast Care, Rochester, New York, United States